CLINICAL TRIAL: NCT07246057
Title: Streamlining Telehealth for Expanded PrEP Utilization Through Community Partnerships (STEP-UP)
Brief Title: Streamlining Telehealth for Expanded PrEP Utilization Through Community Partnerships
Acronym: STEP-UP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Stephen Bonett, Assistant Professor, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R34MH139435 (NIH); 1R34MH139435 (NIH)
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: HIV
Keywords: Pre-exposure prophylaxis; Telehealth; Community-based organizations; Implementation science

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEP-UP Partner Site Model (Experimental): STEP-UP is a partner site model that aims to expand access to telehealth PrEP services for people who could benefit from HIV prevention tools. The first year of the proposed project is dedicated to collaboratively developing and refining the specifics of the STEP-UP model. While the final model will be determined by this formative process, key components will likely include: 1) Establishing a private, on-site space at community-based organizations (CBOs) where clients can engage in telehealth visits with remote PrEP providers; 2) Providing CBOs with the necessary technology and equipment to facilitate telehealth visits; 3) Training CBO staff as Community TelePrEP Navigators to help clients prepare for and follow-up after telehealth appointments, and conduct community-based PrEP education and linkage. Clients referred through the STEP-UP model can schedule appointments with assistance from a Community TelePrEP Navigator or through documented referrals to the self-scheduling tool on the
  Interventions: Behavioral: STEP-UP
- Direct-to-Consumer Telehealth Model (Active Comparator): The existing direct-to-consumer model for telehealth PrEP delivery through the Philadelphia TelePrEP Program. In this model, appointments can be scheduled with assistance from patient navigators and chat operators, or through the self-scheduling tool on the website. This represents the current standard approach for telehealth PrEP service delivery and serves as the comparison group for assessing the preliminary effectiveness of the STEP-UP model.
  Interventions: Behavioral: Philadelphia TelePrEP Program Direct-to-Consumer Model

INTERVENTIONS:
Behavioral: STEP-UP — STEP-UP is a partner site model that aims to expand access to telehealth PrEP services for people who could benefit from HIV prevention tools. The first year of the proposed project is dedicated to collaboratively developing and refining the specifics of the STEP-UP model. While the final model will be determined by this formative process, key components will likely include: 1) Establishing a private, on-site space at community-based organizations (CBOs) where clients can engage in telehealth visits with remote PrEP providers; 2) Providing CBOs with the necessary technology and equipment to facilitate telehealth visits; 3) Training CBO staff as Community TelePrEP Navigators to help clients prepare for and follow-up after telehealth appointments, and conduct community-based PrEP education and linkage. Clients referred through the STEP-UP model can schedule appointments with assistance from a Community TelePrEP Navigator or through documented referrals to the self-scheduling tool on the
  Other Names: Streamlining Telehealth for Expanded PrEP Utilization through community Partnerships
  Arms: STEP-UP Partner Site Model
Behavioral: Philadelphia TelePrEP Program Direct-to-Consumer Model — The existing direct-to-consumer model for telehealth PrEP delivery through the Philadelphia TelePrEP Program. In this model, appointments can be scheduled with assistance from patient navigators and chat operators, or through the self-scheduling tool on the website. This represents the current standard approach for telehealth PrEP service delivery and serves as the comparison group for assessing the preliminary effectiveness of the STEP-UP model.
  Arms: Direct-to-Consumer Telehealth Model

SUMMARY:
The goal of this study is to learn if STEP-UP (Streamlining Telehealth for Expanded PrEP Utilization through community Partnerships) works to expand access to PrEP for people who could benefit from HIV prevention tools. STEP-UP is an innovative model for PrEP delivery that positions community-based organizations (CBOs) as hubs for PrEP access. STEP-UP builds on the established trust, community expertise, and comprehensive services of CBOs serving individuals who could benefit from HIV prevention tools, integrating telehealth PrEP delivery into their existing infrastructure through partnership with a local telehealth PrEP program. By enabling CBOs to offer telePrEP navigation within their array of health and social services, STEP-UP creates accessible, comprehensive care centers that address barriers to PrEP access faced by individuals who could benefit from HIV prevention tools. The main questions it aims to answer are:

1. Is STEP-UP acceptable and feasible to implement in community settings?
2. Does STEP-UP increase PrEP prescription rates compared to the existing direct-to-consumer telehealth model?

Researchers will compare people who receive telehealth PrEP services through STEP-UP at community-based organizations to those who access telehealth PrEP through the existing direct-to-consumer telehealth model. Some participants will:

1. Complete surveys about their experiences with the program
2. Participate in an interview to share their perspectives and feedback about the program.

DETAILED DESCRIPTION:
HIV remains a significant public health challenge in the United States, with new diagnoses concentrated among key populations that continue to experience higher rates relative to the general population. Pre-exposure prophylaxis (PrEP) is a highly effective biomedical prevention tool, but its adoption has been hindered by barriers to healthcare access, resulting in suboptimal utilization rates and limiting its potential to reduce HIV incidence. Telehealth delivery of PrEP (telePrEP) has emerged as a promising strategy for expanding access by overcoming barriers such as transportation, scheduling, and privacy concerns. However, evidence suggests that its reach to individuals at elevated risk for HIV acquisition remains limited, likely due to limitations in technology access, awareness of PrEP, and trust in healthcare systems. To address these challenges, the investigators propose to develop and evaluate STEP-UP (Streamlining Telehealth for Expanded PrEP Utilization through community Partnerships), an innovative model that positions community-based organizations (CBOs) as hubs for PrEP access. STEP-UP builds on the established trust, community expertise, and comprehensive services of CBOs serving people who could benefit from HIV prevention tools, integrating telehealth PrEP delivery into their existing infrastructure through partnership with a local telePrEP program. By enabling CBOs to offer telePrEP navigation within their array of health and social services, STEP-UP creates accessible, comprehensive care centers that address barriers to PrEP access faced by people who could benefit from HIV prevention tools. Through a 3-year observational hybrid implementation-effectiveness pilot study, the investigators aim to: (1) identify multi-level determinants of STEP-UP implementation and collaboratively develop protocols through client interviews (n=20) and workflow observations; (2) characterize implementation outcomes including acceptability, cost, and reach to people who could benefit from HIV prevention tools through surveys with STEP-UP participants (n=50), implementation interviews with stakeholders (n=12), and analysis of program data from CBO partner sites; and (3) assess the preliminary effectiveness of STEP-UP in increasing PrEP prescription rates compared to the current direct-to-consumer model through analysis of program data from the telePrEP program.

ELIGIBILITY:
Inclusion -

Client Interviews:

1. At least 16 years of age or older
2. Have received services or participated in programming at a partner CBO in the past 12 months
3. Currently live in the Philadelphia metropolitan area
4. Able to provide informed consent

Staff Interviews:

1. At least 18 years of age or older
2. Currently employed at Philadelphia telePrEP Program or a partner CBO
3. Serve in a client-facing role (e.g., outreach specialists) or leadership position (e.g., program coordinators) at one of the aforementioned organizations
4. Have been in their current role for at least 6 months
5. Able to provide informed consent

Client Surveys:

1. At least 16 years of age or older
2. Have engaged with a Community TelePrEP Navigator through a partner site CBO to schedule a telehealth appointment with a PrEP provider
3. Currently live in the Philadelphia metropolitan area
4. Able to provide informed consent

Exclusion-

1. Under 16 years of age (clients) or under 18 years of age (staff)
2. Do not currently live in the Philadelphia metropolitan area
3. Unable to provide informed consent due to cognitive impairment or other factors
4. Individuals who pose a safety risk to research staff or other participants
5. Clients currently living with HIV

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
PrEP Prescription Rate | 18-month pilot period
  The proportion of clients who receive a PrEP prescription among those who schedule a telehealth appointment with a PrEP provider. This measure will be compared between clients referred through the STEP-UP partner site model and those engaged through the existing direct-to-client telehealth model.

SECONDARY OUTCOMES:
Acceptability of STEP-UP | Immediately after initial engagement with Community TelePrEP Navigator and 2-4 weeks after initial engagement
  Client-reported acceptability of the STEP-UP model measured using the 8-item Client Satisfaction Questionnaire. The total scores for this scale range from 8 to 32, with the higher number indicating greater acceptability. This validated measure assesses overall satisfaction with services received.
Usability of STEP-UP | Immediately after initial engagement with Community TelePrEP Navigator and 2-4 weeks after initial engagement
  Client-reported usability of the STEP-UP model measured using the 2-item Usability Metric for User Experience LITE scale. The total scores for this scale range from 2 to 14, with the higher number indicating greater usability. This validated measure assesses ease of use of the telehealth PrEP navigation services.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data generated by this study will be archived in the National Institute of Mental Health Data Archive (NDA). The NDA is a secure, federated data repository that provides infrastructure for sharing research data, tools, methods, and analyses enabling collaborative science and discovery. All direct identifiers will be removed and indirect identifiers will be generalized to prevent re-identification.
Time Frame: The investigators will submit our data to the NDA as soon as possible after study completion and data cleaning, and no later than upon publication of the primary study findings. The investigators will protect the rights and privacy of human subjects who participate in sponsored research by redacting all identifiers, and adopting other strategies to minimize risks of unauthorized disclosure of personal identifiers. The NDA will determine the duration of data preservation. To date, the NDA has not removed any data that has been deposited in the repository.
Access Criteria: Researchers interested in accessing the data will follow the NDA standard access procedures. The NDA Data Access Committee will review all requests and determine which ones to approve. If granted access, researchers will have permission to use the data for one year, with the option to renew their access request.